CLINICAL TRIAL: NCT05442424
Title: Keiki (Pediatric) Produce Prescription (KPRx) Program: Quantifying Health Impacts of Healthy Food Prescriptions on Food Security, Health, and Microbiome and Parent-Child Dyads in Hawaii
Brief Title: Keiki (Pediatric) Produce Prescription (KPRx) Program Hawaii
Acronym: KPRxHawaii
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Precision Nutrition KPRx; 1P20GM139753-01A1 (NIH)
Record Dates: First submitted 2022-06-09; First posted 2022-07-05 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Malnutrition, Child; Obesity; Food Selection; Nutrition Poor
Keywords: food insecurity; obesity; nutrition
MeSH Terms: conditions — Child Nutrition Disorders; Obesity; Food Preferences; Malnutrition

STUDY DESIGN:
Intervention Model Description: Randomized control trial, 100 parent-child dyads will receive either $60 per month in vouchers to purchase fresh fruits and vegetables from the community farmers market for 6 months (intervention) or $360 gift certificate to the local grocery store.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Produce Vouchers (Experimental): Half of parent-child dyads will receive $60 per month for 6 months, to purchase fresh fruits and vegetables from a local farmers' market.
  Interventions: Behavioral: Produce Voucher
- Wait-List Control (Active Comparator): Half of parent-child dyads will be placed on a 6 month wait list and will receive $60 per month for 6 months, to purchase fresh fruits and vegetables from a local farmers' market, after completing the 6 month waiting period and follow up data collection.
  Interventions: Behavioral: Wait-List Control

INTERVENTIONS:
Behavioral: Produce Voucher — see arm/group description
  Arms: Produce Vouchers
Behavioral: Wait-List Control — see arm/group description
  Arms: Wait-List Control

SUMMARY:
Children living in food-insecure homes, defined as at some time during the last year their household not having enough food, money, or resources to feed the family experience low intake of fresh fruits and vegetables (FV), and a trajectory for increased risk of obesity and chronic diseases in adulthood. In Hawai'i, a higher proportion of Native Hawaiian (NH) and other Pacific Islander (OPI) children live in food-insecure households when compared with the state average (30% and 50%, respectively vs. 18%) and NHOPI adults suffer disproportionately from chronic disease. Produce prescription programs, provide vouchers to individuals to purchase fresh FV, are promising strategies to improve diet quality and reduce chronic disease risk among food insecure populations. The long-term objective of this research is to reduce nutrition-related health disparities via clinical-community based programming. The Keiki (child) Produce Prescription (KPRx) program was developed and implemented by enlisting University and community researchers and health care providers at the Waianae Coast Comprehensive Health Center (WCCHC). The current study builds on the community-academic partnership to achieve the following specific aim, to measure effectiveness of the KPRx on FV intake, gut microbiome composition, and health related biomarkers in 100 parent-child dyads in the context of household food insecurity from a predominantly NHOPI community in Hawai'i. A community based participatory research approach to carry out a randomized controlled trial that measures the effect of the KPRx on child diet and microbiome, and parent/caregiver diet and health-related biomarkers on 100 parent-child dyads in the context of household food insecurity will be conducted. The community-informed research study will provide data to inform local and state healthcare and nutrition assistance programming policies aimed at reducing food insecurity and health disparities among NHOPI and minority populations.

DETAILED DESCRIPTION:
This Randomized Clinical Trial will recruit and enroll 100 parent-child dyads into 1 of 2 groups, intervention and delayed intervention (control). Participants will be recruited from the Waianae Coast Comprehensive Health Center (WCCHC) pediatrics clinic by pediatricians and primary care providers. Pediatricians will notify study staff of interested participants through the electronic medical record. Study staff will contact participants to share more study information and schedule a time for enrollment.

The first enrollment appointment will take place via phone. Prior to the appointment participants will be sent the informed consent and baseline study surveys. These will be administered by a trained researcher over the phone. Baseline survey responses will be recorded in RedCAP. Participants will then be instructed to pick up the stool collection kits at WCCHC and scheduled to come in for an in-person specimen drop off and further data collection. At this second appointment participants will drop off stool samples (one for parent and one for child). Parents and children will also be asked to complete a reflective spectroscopy test (VeggieMeter) and parents' will complete the following measures: blood pressure, weight, finger stick lipids (AccuCheck) and hemoglobin A1c (A1C now). Trained staff will follow the study procedure for conducting the finger stick to obtain the blood sample and follow all safety protocols for handling blood. Measures will be recorded in RedCap by study staff.

Participants will be notified of randomization group (intervention or control). Intervention participants will receive their first $60 voucher for fresh fruits and vegetables and be instructed on how to redeem it at the farmers market. Control participants will receive a $50 gift card to a local store.

Intervention participants will receive $60 each month for 6 months of the intervention. These funds will be uploaded onto a gift card. Participants will be able to use the gift card at produce vendors at the farmers' market. The funds will expire each month.

Six months after enrollment, all participants will be schedule to complete the baseline assessments again. This will include the survey, stool samples, and Veggie Meter reading for parents and children; and the lipids, A1c, blood pressure, and weight for parents. Intervention group participants will receive a $50 gift card to a local store. Control group participants will receive their first of six $60 vouchers for fresh fruits and vegetables and be instructed on how to redeem it at the farmers market.

Baseline and 6 month Survey questions will include the Current Population Survey's food security questions and the Dietary Screener Questionnaire for assessing fruit and vegetable consumption.

ELIGIBILITY:
Inclusion Criteria:

* patient of the Waianae Coast Comprehensive Health Center (WCCHC) Pediatric Clinic
* 2 to 8 years of age
* positive screen for food insecurity using a validated two-question tool,44 and/or has overweight or obese, BMI ≥ 85th percentile, measurement recorded in Electronic Medical Record (EMR) on day of clinic visit when recruitment occurs)
* resides with the parent on the Wai'anae Coast of O'ahu
* English-speaking.

Exclusion Criteria:

* individuals > 8 years of age
* children who are not WCCHC pediatric patients
* children who do not experience food security
* non-English speaking children
* children living outside of the Wai'anae Coast of O'ahu

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 170 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Change in Child Fruit and Vegetable Intake at six months | baseline and 6 months from enrollment
  daily fruit and vegetable intake (servings per day) of child measured with (Dietary Screener Questionnaire (DSQ) 2009-10. National Cancer Institute). Unit of measure will be the change in number of servings of fruits and vegetables consumed per day by child.

SECONDARY OUTCOMES:
Change in Parent- Blood Pressure at six months | baseline and 6 months from enrollment
  systolic and diastolic blood pressure
Change in Parent- Lipids at six months | baseline and 6 months from enrollment
  Total cholesterol, HDL and LDL cholesterol
Change in Parents- Glucose Control | baseline and 6 months from enrollment
  Hemoglobin A1c
Change in Household food security status | baseline and 6 months from enrollment
  food security measured with Food Security in the United States: Current Population Survey. United States Department of Agriculture Economic Research Service. Unit of measure is the change in percentage of households who are food secure, have low food security, and very low food security.
Change in Parent Fruit and Vegetable Intake | baseline and 6 months from enrollment
  daily fruit and vegetable intake (servings per day) of parent/caregiver measured with Dietary Screener Questionnaire (DSQ) 2009-10. National Cancer Institute. Unit of measure will be change in the number of servings of fruits and vegetables consumed per day by parent/caregiver
Change in Gut Microbiome- Parent | baseline and 6 months from enrollment
  Parents' abundance and richness of the gut microbiome, α-diversity, Firmicutes to Bacteroidetes ratio, and the relative abundance of each member of the microbial communities from phyla to species level
Change in Gut Microbiome- Child | baseline and 6 months from enrollment
  Child's abundance and richness of the gut microbiome, α-diversity, Firmicutes to Bacteroidetes ratio, and the relative abundance of each member of the microbial communities from phyla to species level

CONTACTS AND LOCATIONS:
Overall Officials: Marla Berry, PhD, Study Director — University of Hawaii at Manoa
Locations (1):
- University of Hawaii at Manoa, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No